CLINICAL TRIAL: NCT03206463
Title: Cognitive and Psychophysiological Effects of Delta-9-Tetrahydrocannabinol in Bipolar Disorder
Acronym: THC-BD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Feasibility pilot was completed
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2000020272
Record Dates: First submitted 2017-06-19; First posted 2017-07-02 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Delta-9-Tetrahydroncannabinol; Bipolar Disorder; Healthy Controls
MeSH Terms: conditions — Bipolar Disorder | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: The study is a double-blind, randomized, placebo-controlled, crossover laboratory evaluation of the acute subjective, cognitive and psychophysiological effects of 2 mg and 4 mg inhaled THC in Healthy Control individuals and individuals with euthymic Bipolar Disorder.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active 4 mg inhaled THC (Experimental): Subject will have 1/3 chance of receiving 4 mg THC administered through a vaporizer, over approximately 20 minutes, followed by approximately 45 minutes of neuropsychological and physiological testing.
  Interventions: Drug: 4 mg Delta-9-THC
- Active 2 mg inhaled THC (Experimental): Subject will have 1/3 chance of receiving 2 mg THC administered through a vaporizer, over approximately 20 minutes, followed by approximately 45 minutes of neuropsychological and physiological testing.
  Interventions: Drug: 2 mg Delta-9-THC
- Placebo (Placebo Comparator): Subject will have 1/3 chance of receiving the inhaled placebo condition administered through a vaporizer, over approximately 20 minutes, followed by approximately 45 minutes of neuropsychological and physiological testing. The placebo condition will include no active cannabinoids.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4 mg Delta-9-THC — Subject will have 1/3 chance of receiving 4 mg THC administered through a vaporizer, over approximately 20 minutes, followed by approximately 45 minutes of neuropsychological and physiological testing.
  Arms: Active 4 mg inhaled THC
Drug: Placebo — Subject will have 1/3 chance of receiving the inhaled placebo condition administered through a vaporizer, over approximately 20 minutes, followed by approximately 45 minutes of neuropsychological and physiological testing. The placebo condition will include no active cannabinoids.
  Arms: Placebo
Drug: 2 mg Delta-9-THC — Subject will have 1/3 chance of receiving 2 mg THC administered through a vaporizer, over approximately 20 minutes, followed by approximately 45 minutes of neuropsychological and physiological testing.
  Arms: Active 2 mg inhaled THC

SUMMARY:
The overarching goal of this study is to characterize the acute cognitive and psychophysiological effects of the main psychoactive constituent of cannabis, 9-delta-tetrahydrocannabinol (THC) in individuals with euthymic bipolar disorder (BD), and to begin probing the mechanisms that may underlie its effects in this illness.

This study is expected to contribute to a better characterization of specific effects of THC in individuals with BD compared to healthy controls (HC).

DETAILED DESCRIPTION:
To compare the dose related acute effects of inhaled THC, administered through a vaporizer over approximately 20 minutes, between HC and euthymic BD individuals (referred to as eBD) on a range of subjective and objective parameters as described below:

Primary Aims:

* Verbal memory, measured by a modified computer version of the Rey Auditory Verbal Learning Test (RAVLT) and/or the CogState battery, administered while EEG data is collected.
* Executive functioning measured by the CogState battery and/or Trails Making Test-Part B.

Secondary Aims:

* Attention, measured by the Continuous Performance Test-Identical Pairs (CPT-IP).
* Working memory, measured by the Wechsler Memory Scale-3 Letter-Number Sequencing.
* Mood, measured by the Profile of Mood States (POMS).
* Psychotic-type experiences, measured by the Psychotomimetic States Inventory (PSI) and/or the Clinician Administered Dissociative Symptoms Scale (CADSS).
* Anxiety symptoms, measured by the Visual Analog Scale for Anxiety (VAS-A).
* Impulsivity, measured by the Balloon Analogue Risk Task (BART).

Exploratory aims:

•Serum prolactin, serum ACTH, serum cortisol and serum endocannabinoid levels.

ELIGIBILITY:
Inclusion Criteria for individuals with Bipolar Disorder (BD)

1. Men and women aged 18-55 years (extremes included).
2. Able to provide informed consent in English.
3. A diagnosis of BD type I or BD type II and good physical health.
4. Current euthymic state for at least 4 weeks.

Inclusion Criteria for Healthy Control (HC) individuals:

1. Men and women aged approximately 18-55 years (extremes included).
2. Able to provide informed consent in English.
3. No psychiatric diagnoses and in good physical health.

General exclusion criteria:

1. Cannabis naïve
2. Unwillingness to remain alcohol-free, cannabis-free for at least 1 week (in infrequent cannabis users) prior to each test day.
3. Evidence of a hearing deficit.
4. IQ less than 80.
5. Positive pregnancy test, lactation, and refusal to practice birth control.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Change in Verbal memory | baseline and +35 mins after drug administration
  Verbal memory will be measured by a modified computer version of the Rey Auditory Verbal Learning Test (RAVLT) and/or the CogState battery, administered while EEG data is collected.
Change in Executive functioning | baseline and +35 mins after drug administration
  Executive functioning will be measured by the CogState battery and/or Trails Making Test-Part B.

SECONDARY OUTCOMES:
Attention | baseline and +35 mins after drug administration
  Attention will be measured by the Continuous Performance Test-Identical Pairs (CPT-IP).
Working memory | baseline, +35 mins after drug administration, +90 mins after drug administration and +210 mins after drug administration
  Working memory will be tested by the Wechsler Memory Scale-3 Letter-Number Sequencing.
Mood | baseline and +20 mins after drug administration, +90 mins after drug administration and +210 mins after drug administration
  Mood will be measured by the Profile of Mood States (POMS).
Psychotic-type experiences | baseline and +20 mins after drug administration, +90 mins after drug administration and +210 mins after drug administration
  Psychotic-type experiences will be measured by the Psychotomimetic States Inventory (PSI) and/or the Clinician Administered Dissociative Symptoms Scale (CADSS).
Anxiety symptoms | baseline and +20 mins after drug administration, +90 mins after drug administration and +210 mins after drug administration
  Anxiety symptoms will be measured by the Visual Analog Scale for Anxiety (VAS-A).
Impulsivity | baseline, +35 mins after drug administration, +90 mins after drug administration and +210 mins after drug administration
  Impulsivity will be measured by the Balloon Analogue Risk Task (BART).

OTHER OUTCOMES:
Blood serum hormonal levels • Serum prolactin, serum ACTH, serum cortisol and serum endocannabinoid levels. • Serum prolactin, serum ACTH, serum cortisol and serum endocannabinoid levels. | baseline, +20 mins after drug administration, +30 mins after drug administration, +60 mins after drug administration, +90 mins after drug administration, +150 mins after drug administration, +210 mins after drug administration
  As an exploratory aim, serum prolactin (ng/mL), serum ACTH (pg/ml), and serum cortisol (μg/dL) levels will be measured to provide an objective measure of THC effects on the hypothalamic pituitary adrenal (HPA) axis.
Blood serum THC and metabolite levels (ng/ml) | baseline, +20 mins after drug administration, +30 mins after drug administration, +60 mins after drug administration, +90 mins after drug administration, +150 mins after drug administration, +210 mins after drug administration
  Blood levels of THC and both its active and inactive metabolites will be assayed to explore the gender related differences in the metabolism of THC.
Blood pressure | baseline, -60 mins before drug administration, +2, +4, +6, +8,+10, +20, +30, +35, +40, +45, +50, +60, +90, +150, +210 mins after drug administration.
  Blood pressure (mmHg) will be assessed as part of the medical monitoring of the subjects
Pulse | baseline, -60 mins before drug administration, +2, +4, +6, +8,+10, +20, +30, +35, +40, +45, +50, +60, +90, +150, +210 mins after drug administration.
  Pulse (beats per min) will be assessed as part of the medical monitoring of the subjects
Genetics | Only on 1st test day
  Blood samples for DNA extraction will be collected to examine whether any of the genes implicated in cognition in the response to cannabinoids (e.g., COMT, CNR1, FAAH, BDNF) modify the effects of THC.

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, MD, Principal Investigator — Yale University
Locations (1):
- Biological Studies Unit, VA Connecticut Healthcare System, West Haven, Connecticut, United States